CLINICAL TRIAL: NCT03307499
Title: Post-market, Prospective Evaluation of Human Placental Membrane Tissue Used as an Adjunct for Foot and Ankle Tendon Surgery in Patients With Chronic Tendinopathy
Brief Title: NeoPatch Used as Adjunct in Foot and Ankle Tendon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPM1701.000-M
Record Dates: First submitted 2017-09-12; First posted 2017-10-11 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Tendinopathy; Tendon Tear; Tendon Injuries; Foot Ankle Injuries
MeSH Terms: conditions — Tendinopathy; Tendon Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): NeoPatch
  Interventions: Other: NeoPatch

INTERVENTIONS:
Other: NeoPatch — NeoPatch as an adjunct to foot and ankle tendon revision/repair surgery

SUMMARY:
This study is a prospective, single center, postmarket study to evaluate the safety and effectiveness of NeoPatch used as a tissue cover in foot and ankle tendon revision and repair surgery.

DETAILED DESCRIPTION:
This study is a prospective, single center, postmarket study to evaluate the safety and effectiveness of NeoPatch used as a tissue cover for chronically injured tendons requiring surgical revision. NeoPatch is a tissue covering derived from terminally sterilized, dehydrated human placental membrane tissue comprised of both amnion and chorion. Candidates for this study are patients presenting with chronic tendon pain that are being evaluated for primary tendon revision surgery following failure of standard of care or immediate need for surgery, as determined by the investigator. Consented patients will receive NeoPatch as an adjunct to their foot or ankle tendon revision; NeoPatch will be wrapped around the tendon immediately prior to closure. The study will be divided into two phases: Screening and Follow-up. The study will include prospective patient evaluations at scheduled clinic visits and ultrasound appointments for a maximum of 12 visits over 12 months. Patient history, medications, self-reported pain, tendon status, and adverse events will be collected on all patients consented and enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tendinopathy requiring surgical revision in the opinion of the Investigator as defined in Appendix G.
* Intention to schedule surgical revision.

  ≥ 18 years.
* Free from clinical signs of infection at time of screening and at time of surgical intervention.
* Target tendon is one of the following: Achilles, Extensor Digitorum Longus, Extensor Hallucis Brevis, Extensor Hallucis Longus, Flexor Digitorum Longus, Flexor Hallucis Longus, Tibialis Anterior, Tibialis Posterior, Peroneus Longus, Peroneus Brevis, Peroneus Tertius.
* Able and willing to provide consent and comply with protocol.

Exclusion Criteria:

* History of surgical intervention involving target tendon.
* Tendon injury is acute in nature.
* Current participation in another clinical study.
* Currently receiving radiation or chemotherapy.
* Diagnosis of autoimmune connective tissue disease requiring systemic immunomodulatory therapy; stable NSAID doses for mild rheumatoid arthritis permitted.
* Use of biomedical growth factor within previous 30 days.
* Pregnant or breastfeeding or planning on becoming pregnant or unwilling to use medically acceptable methods of birth control.
* Taking medications considered to be immune system modulators within previous 30 days.
* Patient taking specific Cox-2 inhibitors within previous 30 days.
* Currently being treated with an investigational device or drug (within 3 months prior to surgery).
* Allergy, intolerance or hypersensitivity to any components or packaging of the product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Quantitative ultrasound assessment of post-operative adhesions | Up to 3 weeks, post-op
  Average physical measurement of target tendon adhesions in mm, by ultrasound assessment.
Quantitative ultrasound assessment of post-operative adhesions | Up to 9 weeks, post-op
  Average physical measurement of target tendon adhesions in mm, by ultrasound assessment.
Quantitative ultrasound assessment of post-operative adhesions | Up to 15 weeks, post-op
  Average physical measurement of target tendon adhesions in mm, by ultrasound assessment.
Quantitative ultrasound assessment of post-operative adhesions | Up to 52 weeks, post-op
  Average physical measurement of target tendon adhesions in mm, by ultrasound assessment.
Change in quantitative ultrasound assessment of post-operative adhesions | Through study completion, an average of 1 year
  Average percent change in physical measurement of target tendon adhesions, by ultrasound assessment.
Qualitative ultrasound assessment of post-operative adhesions | Up to 3 weeks, post-op
  Categorical summary of adhesion severity, reported by ultrasound assessment, described as mild, moderate, or severe.
Qualitative ultrasound assessment of post-operative adhesions | Up to 9 weeks, post-op
  Categorical summary of adhesion severity, reported by ultrasound assessment, described as mild, moderate, or severe.
Qualitative ultrasound assessment of post-operative adhesions | Up to 15 weeks, post-op
  Categorical summary of adhesion severity, reported by ultrasound assessment, described as mild, moderate, or severe.
Qualitative ultrasound assessment of post-operative adhesions | Up to 52 weeks, post-op
  Categorical summary of adhesion severity, reported by ultrasound assessment, described as mild, moderate, or severe.

SECONDARY OUTCOMES:
VAS Average Pain Score | Up to 1 year, post-op
  Average self-reported pain experienced on average
VAS Current Pain Score | Up to 1 year, post-op
  Average self-reported pain experienced at time of assessment (current)
Change in VAS Average Pain Score | Through study completion, an average of 1 year
  Average change in self-reported average pain from baseline (screening) to last follow-up visit.
Change in VAS Current Pain Score | Through study completion, an average of 1 year
  Average change in self-reported current pain from baseline (screening) to last follow-up visit.
AOFAS Foot and Ankle Function Score | Up to 24 weeks, post-op
  Average AOFAS score
AOFAS Foot and Ankle Function Score | Up to 52 weeks, post-op
  Average AOFAS score
Change in AOFAS Foot and Ankle Function Score | Up to 24 weeks, post-op
  Average AOFAS score change between baseline (Screening) and Visit 7
Change in AOFAS Foot and Ankle Function Score | Up to 52 weeks, post-op
  Average AOFAS score change between baseline (Screening) and Visit 8
Use of Analgesics | Up to 52 weeks, post-op
  Percentage of patients on analgesics, including NSAIDs and narcotics, for the treatment of their target tendon pain.
Change in the Use of Analgesics | Through study completion, an average of 1 year
  Percent change of patients on analgesics, including NSAIDs and narcotics, for the treatment of their target tendon pain.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Pacaccio, DPM, Principal Investigator — Advanced Foot and Ankle Surgeons
Locations (1):
- Advanced Foot and Ankle Surgeons, Sycamore, Illinois, United States